CLINICAL TRIAL: NCT06145009
Title: Time Restricted Eating, Eating Behaviors, and Cardiometabolic Risk in Emerging Adult Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Carly R Pacanowski, Associate Professor, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2089190-1
Record Dates: First submitted 2023-10-17; First posted 2023-11-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Time Restricted Eating; Eating Behavior; Diet, Healthy; Nutrition, Healthy
MeSH Terms: conditions — Intermittent Fasting; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time Restricted Eating (Experimental): Participants will limit their eating (all food and caloric beverages) to an eating window of 10 hours per day for 4 weeks. The eating window must end by 8pm. Water and non-caloric beverages are allowed outside of the eating window. No other changes are required to the types or total amount of food eaten.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Limit food intake to 10 hours per day as described in the experimental arm section.
  Other Names: Time restricted feeding; Intermittent fasting; Meal timing

SUMMARY:
The purpose of this study is to assess how time restricted eating interventions impact eating behaviors, diet quality, and body composition in women ages 20-29 years. Participants will be asked to limit all food and drinks (except water and some non-caloric beverages) to a 10-hour period during the day for four weeks. Participants will follow their usual eating and activity patterns for one week before starting, and follow whatever eating pattern they want for 4 weeks after finishing.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Own a smartphone
* BMI ≥ 20 kg/m2
* Usual eating window ≥ 12 hours with the last eating occasion after 8pm on the majority of days
* Have at least a moderate baseline level of dietary restraint

Exclusion Criteria:

* Shift workers
* Being pregnant, nursing, or planning to become pregnant in the next 6 months
* Having a past or current eating disorder diagnosis
* Having a chronic medical condition (including diabetes, heart, kidney, or thyroid disease) or a condition that requires therapeutic diet or specified meal timing

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — People who identify as a woman are eligible.
Enrollment: 36 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Emotional Eating | 3 time points: baseline, end of 4-week intervention, end of 4-week follow up
  Dutch Eating Behavior Questionnaire: Emotional Eating Subscale. This subscale is scored from 1-5, with higher scores indicating higher emotional eating.
External Eating | 3 time points: baseline, end of 4-week intervention, end of 4-week follow up
  Dutch Eating Behavior Questionnaire: External Eating Subscale. This subscale is scored from 1-5, with higher scores indicating higher external eating.
Eating in the Absence of Hunger | Baseline week, weeks 1 and 4 of intervention, weeks 1 and 4 of follow up
  Assessed through surveys sent 5x/day asking about if food was eaten and why.

SECONDARY OUTCOMES:
Diet Quality | 3 time points: baseline, end of 4-week intervention, end of 4-week follow up
  Healthy Eating Index, calculated from 3-day food records. The Healthy Eating Index is scored from 0-100, with higher scores indicating higher diet quality.
Body composition (total percent body fat) | Baseline and end of 4-week intervention
  Percent body fat measured by DXA
Body composition (visceral fat) | Baseline and end of 4-week intervention
  Visceral fat measured by DXA
Body weight | 3 time points: baseline, end of 4-week intervention, end of 4-week follow up
  Total body weight

OTHER OUTCOMES:
Participant experience | End of 9-week study (following 1-week baseline, 4-week intervention, and 4-week follow up)
  Qualitative interview to glean information on participants' subjective experience of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carly Pacanowski, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States